CLINICAL TRIAL: NCT00377988
Title: The Risk of Venous Thromboembolism, Myocardial Infarction, and Ischemic Stroke Among Women Using the Transdermal Contraceptive System Compared With Women Using Norgestimate-containing Oral Contraceptives With 35 mcg Ethinyl Estradiol
Brief Title: A Postmarketing Study of the Risk of Venous Thromboembolism (Blood Clots), Myocardial Infarction (Heart Attacks), and Stroke Among Women Using ORTHO EVRA (Norelgestromin and Ethinyl Estradiol Contraceptive Patch) Compared With Women Who Take Oral Contraceptives for Birth Control
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR012022; EVRA-13-MAGNIFI
Record Dates: First submitted 2006-09-15; First posted 2006-09-19 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Contraception; Female Contraception
Keywords: Contraception; Hormonal contraception; Oral contraception; Ethinyl estradiol; Progestin; Transdermal; Thrombosis; Venous thromboembolism
MeSH Terms: conditions — Thrombosis; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- 001: Transdermal Contraceptive System In each 4-week period exposed subjects will wear a transdermal patch containing 6 mg norelgestromin and 0.75 mg EE worn for each of 3 consecutive weeks with no patch the 4th week.
  Interventions: Drug: Transdermal Contraceptive System
- 002: Norgestimate-containing oral contraceptives with EE NGM-OCs with 34 mcg of EE taken during each 4 week period for 21 consecutive days then no pill or a drug-free pill 7 days.
  Interventions: Drug: Norgestimate-containing oral contraceptives with EE

INTERVENTIONS:
Drug: Transdermal Contraceptive System — In each 4-week period, exposed subjects will wear a transdermal patch containing 6 mg norelgestromin and 0.75 mg EE worn for each of 3 consecutive weeks with no patch the 4th week.
  Groups: 001
Drug: Norgestimate-containing oral contraceptives with EE — NGM-OCs with 34 mcg of EE taken during each 4 week period for 21 consecutive days, then no pill or a drug-free pill 7 days.
  Groups: 002

SUMMARY:
The purpose of the study is to use data from a health care information database to assess the risk of venous thromboembolism (blood clots), myocardial infarction (heart attacks), and stroke among women using a transdermal contraceptive system (ORTHO EVRA) for birth control compared with women using norgestimate-containing oral contraceptives with 35 mcg ethinyl estradiol.

DETAILED DESCRIPTION:
ORTHO EVRA (norelgestromin and ethinyl estradiol) is a once-a-week transdermal contraceptive (birth control) system where a small square-shaped patch is worn on the body and hormones from the patch are absorbed transdermally (through the skin) to help prevent pregnancy. This is an observational case-control study that will use data provided by a United States health care claims database and the National Death Index (NDI) to assess the risk of venous thromboembolism abbreviated as VTE (includes deep vein thrombosis abbreviated as DVT [a blood clot that forms in one or more of the deep veins of the body, usually the legs] and pulmonary embolism abbreviated as PE [a blood clot in the lungs]), acute myocardial infarction abbreviated as AMI (heart attack), and ischemic stroke (blockage of an artery that supplies blood to the brain) among women using the transdermal contraceptive system, ORTHO EVRA compared with women using norgestimate-containing oral contraceptives (NGM-OCs) with 35 mcg ethinyl estradiol (EE), during the period 01 April 2002 to 31 December 2004 and during an extension period from 01 January 2005 to 31 December 2006. In the extension period of the study (01 January 2005 to 31 December 2006), mortality was added as an endpoint in the study. After obtaining Institutional Review Board (IRB) approval and a waiver of authorization, requests will be made for medical records for all women who have been dispensed at least once with ORTHO EVRA or a NGM-OC and whose health insurance claims are consistent with the occurrence of VTE, AMI, or stroke. The primary outcome measure in the study is AMI and ischemic stroke combined in current and recent users or ORTHO EVRA compared to current and recent users of NGM-OCs with 34 mcg of EE. Observational study - No investigational drug administered. NOTE: The study was conducted in two parts. Study CR014383, NCT00511784, represents the first portion of the study. This study, CR012022, represents the second portion of the extended study.

ELIGIBILITY:
Inclusion Criteria:

* Users of a transdermal contraceptive system or norgestimate-containing oral contraceptives with 35 mcg ethinyl estradiol between April 1, 2002 and December 31, 2006, who are identified in the Ingenix Research Database
* Have complete medical coverage and pharmacy benefits

Exclusion Criteria:

* Have a claim associated with physician services for any of the following: malignancy other than non-melanoma skin cancer
* coagulation defects, history of venous thrombus/embolism, or long-term anticoagulant use
* Chronic inflammatory disease

Ages: 15 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women using a transdermal contraceptive system or NGM-OCs containing 35 mcg EE between April 1, 2002 and December 31, 2006 whose medical records are accessable through research databases in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 423 (Actual)
Dates: Start 2002-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
AMI and ischemic stroke combined in current and recent users or ORTHO EVRA compared to current and recent users of NGM-OCs with 34 mcg of EE. | From 01 April 2002 to 31 December 2004 combined with data from the extension period from 01 January 2005 to 31 December 2006.

SECONDARY OUTCOMES:
AMI in current and recent users or ORTHO EVRA compared to current and recent users of NGM-OCs with 34 mcg of EE. | From 01 April 2002 to 31 December 2006.
Ischemic stroke in current and recent users or ORTHO EVRA compared to current and recent users of NGM-OCs with 34 mcg of EE. | From 01 April 2002 to 31 December 2006.
VTE (a combined outcome of PE and DVT) in current and recent users or ORTHO EVRA compared to current and recent users of NGM-OCs with 34 mcg of EE. | From 01 April 2002 to 31 December 2006.
AMI or ischemic stroke or VTE combined in current and recent users or ORTHO EVRA compared to current and recent users of NGM-OCs with 34 mcg of EE. | From 01 April 2002 to 31 December 2006.
All deaths (identified by the NDI), NDI-identified deaths due to AMI, ischemic stroke or VTE, and NDI-identified deaths due to sudden or unknown causes | From 01 April 2002 to 31 December 2006.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Cole JA, Norman H, Doherty M, Walker AM. Venous thromboembolism, myocardial infarction, and stroke among transdermal contraceptive system users. Obstet Gynecol. 2007 Feb;109(2 Pt 1):339-46. doi: 10.1097/01.AOG.0000250968.82370.04. PMID 17267834
- See also: Myocardial infarction, stroke, and venous thromboembolism among transdermal contraceptive system users — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=738&filename=CR012022_REF1.pdf
- See also: Dore DD, Norman H, Loughlin J, Seeger JD (in press). Extended case-control study results on thromboembolic outcomes among transdermal contraceptive users. Contraception. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=738&filename=CR012022_REF2.pdf
- See also: Myocardial infarction, stroke, and venous thromboembolism among transdermal contraceptive system users — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=738&filename=CR012022_REF3.pdf